CLINICAL TRIAL: NCT07230652
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose- Ascending Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of LPM787000048 Maleate Extended-Release Tablets (LY03020) in Chinese Adult Healthy Subjects and/or Subjects With Stable Schizophrenia
Brief Title: A Phase 1 MAD Study to Evaluate the Safety and Tolerability of LY03020
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03020/CT-CHN-103
Record Dates: First submitted 2025-08-06; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia; Alzheimer's Disease Psychosis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY03020 (Experimental): Subjects will take LY03020 from Day 1 to Day 7
  Interventions: Drug: LY03020
- Placebo (Placebo Comparator): Subjects will take Placebo from Day 1 to Day 7
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03020 — administered orally
  Arms: LY03020
Drug: Placebo — administered orally
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, ascending multiple oral dose study to assess the safety, tolerability, and pharmacokinetics of LY03020 in Chinese healthy adult subjects and/or subjects with stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects

* Subjects sign informed consent voluntarily.
* Male or female aged 18 to 45 years.
* Body weight ≥ 50.0 kg for male and ≥ 45.0 kg for female, and body mass index (BMI) between 18.5 and 26.0 kg/m2 Subjects with Stable Schizophrenia
* Subjects themselves and / or their guardians sign informed consent voluntarily.
* Male or female aged 18 to 60 years.
* Body weight ≥ 50.0 kg for male and ≥ 45.0 kg for female, and body mass index (BMI) between 18.5 and 32.0 kg/m2.
* Subject must meet the DSM-V criteria for a primary diagnosis of schizophrenia. Subject must have a PANSS total score ≤ 80 and CGI-S score ≤ 4 at screening. The condition is stable from 1 month before signing informed consent to baseline.

Exclusion Criteria:

Healthy Subjects

* Subjects have any clinically significant medical condition or chronic disease.
* Subjects have used any of nonprescription drugs within 7 days or prescription drugs within 28 days prior to administration.
* Subjects experienced a history of keratopathy, fundus disease, increased intraocular pressure, or angle-closure glaucoma. Subjects have any abnormal and clinically significant test for ophthalmic examination during screening.
* Subjects with a history of orthostatic hypotension or syncope.
* Subjects with condition that may interfere with the drug absorption, distribution, metabolism and excretion significantly.
* Subjects had a history of surgery within 3 months prior to administration, or had not recovered, or have a surgical plan during the study.
* Subjects have any clinically significant abnormal vital signs, laboratory values, and ECGs.
* Subjects have a history of allergic diseases, or allergic to any substance contained in the formulation
* Subjects have a positive test for HBsAg, HCV-Ab, HIV-Ab, or syphilis antibody. Subjects with Stable Schizophrenia
* According to the DSM-5, there were other mental disorders except schizophrenia within 6 months before screening period.
* Assessed by the investigator as having treatment-resistant schizophrenia; past or current diagnosis of neuroleptic malignant syndrome (NMS); anticipated need for antipsychotic regimen modifications during the study period;
* History of suicide attempts (including actual attempts, interrupted attempts, or failed attempts) or suicidal ideation within the past 6 months, defined as affirmative responses ("yes") to question 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening/baseline;
* Subjects have used monoamine oxidase inhibitors (MAOI) within 28 days or any dietary supplements/traditional Chinese herbal products within 7 days prior to first dosing.
* Glycated hemoglobin (HbA1c) ≥7% at screening/baseline.
* Congenital long QT syndrome; uncontrolled or severe cardiovascular disease, including NYHA class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months prior to screening, or presence of treatment-requiring severe arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) at screening; resting heart rate <50 beats per minute (bpm) at screening/baseline; or QTc >450 ms (male) / QTc >460 ms (female) based on Fridericia's formula-corrected measurements at screening/baseline.
* Subjects experienced a history of keratopathy, fundus disease, increased intraocular pressure, or angle-closure glaucoma. Subjects have any abnormal and clinically significant test for ophthalmic examination during screening.
* Subjects with a history of orthostatic hypotension or syncope.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs). | up to Day 11

SECONDARY OUTCOMES:
Number of participants with clinical laboratory assessment abnormalities. | up to Day 11
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) at Day 11 of subjects with stable schizophrenia | up to Day 11
  The total score range is 30 to 210.A higher score is associated with greater illness severity.
Change from Baseline in Columbia - Suicide Severity Rating Scale (C-SSRS) at Day 11 of subjects with stable schizophrenia | up to Day 11
  This scale is divided into three parts, which are evaluated suicidal ideation(5 items [yes/no])，intensity of ideation (5 items on 5-point scales; scores range from 0 to 25 with higher scores indicating more intense suicidal ideation),and suicide behavior(actual attempt,interrupted attempt,aborted attempt, preparatory acts or behavior).
Change from Baseline in Barnes Akathisia Rating Scale (BARS) at Day4 and Day 11 of subjects with stable schizophrenia | up to Day 11
  The total score range is 0 to 14.A higher score is associated with greater illness severity.
Change from Baseline in Simpson-Angus Scale (SAS) at Day4 and Day 11 of subjects with stable schizophrenia | up to Day 11
  This scale consists of 10 items, and each question is scored from 0 to 4 points. The Total score range is 0 to 40.A higher score is associated with greater illness severity.
Maximum observed concentration at steady state (Cmax,ss) of LPM787000048 in plasma | up to Day 11
Minimum observed concentration at steady state (Cmin,ss) of LPM787000048 in plasma | up to Day 11
Area under the concentration- time curve during the dosing interval at steady state (AUC0-τ,ss) of LPM787000048 in plasma | up to Day 11
Area under the concentration-time curve from time zero extrapolated to infinity at steady state (AUC0-∞,ss) of LPM787000048 in plasma | up to Day 11
Time to maximum observed concentration at steady (Tmax,ss) state of LPM787000048 in plasma | up to Day 11
Apparent terminal elimination half-life (t1/2) of LPM787000048 in plasma | up to Day 11
AUC Accumulation Ratio (Ra(AUC)) of LPM787000048 in plasma | up to Day 11
Cmax Accumulation Ratio (Ra(Cmax)) of LPM787000048 in plasma | up to Day 11
Number of participants with vital sign abnormalities. | up to Day 11
Number of participants with 12-lead electrocardiogram abnormalities (ECGs). | up to Day 11
Number of participants with ophthalmic examination abnormalities. | up to Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing AnDing Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No